CLINICAL TRIAL: NCT00400582
Title: Effect of ACE Inhibitor Plus High Dose Candesartan on BNP and Inflammation in Patients With LV Dysfunction: Impact of Renin-angiotensin-aldosterone System Genetic Polymorphisms
Brief Title: A Pharmacogenomic Study of Candesartan in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Michel White, Montreal Heart Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHI 06-890; D2454L00003
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Gene polymorphism; Candesartan; ACE inhibitors; BNP; Pharmacogenomics
MeSH Terms: conditions — Heart Failure | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Candesartan up to 32 mg daily — Candesartan 4 to 32 mg daily
  Other Names: Atacand

SUMMARY:
The purpose of this study is to evaluate the impact of genetic variations on the response to candesartan in patients with heart failure who are already treated with an ACE inhibitor.

ELIGIBILITY:
Principal Inclusion Criteria:

1. Male or female > or = 18 years old.
2. Symptomatic CHF corresponding to NYHA class II-IV symptoms for at least 4 weeks prior randomization.
3. LVEF < or = 40%
4. Treatment with an optimal and stable dose of ACE inhibitor for at least 4 weeks prior to enrolment in the study.

Principal Exclusion Criteria:

1. Treatment with an ARB within 8 weeks prior to randomization.
2. Known hypersensitivity to ARBs or ACE inhibitors.
3. Creatinine clearance < 30 ml/min or serum creatinine > 221
4. Current serum potassium > or = 5.0 mmol/L or a history of marked ACE inhibitor or ARB induced hyperkalemia.
5. Known bilateral renal artery stenosis.
6. Current symptomatic hypotension and/or systolic B.P. < 90 mmHg.
7. Decompensated heart failure described as hospitalization or I.V. administration of medication in emergency room or heart failure clinic within 4 weeks
8. Stroke, acute coronary syndrome, PCI within the last 4 weeks before randomization.
9. Connective tissue disease or chronic inflammatory condition
10. Acute inflammatory process such as an infection or gout attack in the last 2 weeks.
11. Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
BNP and NT-proBNP | 16 weeks

SECONDARY OUTCOMES:
Blood pressure | 16 weeks
CRP | 16 weeks
Renin | 16 weeks
Aldosterone | 16 weeks
Insulin resistance/ glucose | 16 weeks
NYHA functional class | 16 weeks
Tolerability | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michel White, MD, Principal Investigator — Montreal Heart Institute; Simon de Denus, B. Pharm, MSc,PhD, Principal Investigator — Montreal Heart Institute/ Faculty of Pharmacy, University of Montreal
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] de Denus S, Dube MP, Fouodjio R, Huynh T, LeBlanc MH, Lepage S, Sheppard R, Giannetti N, Lavoie J, Mansour A, Provost S, Normand V, Mongrain I, Langlois M, O'Meara E, Ducharme A, Racine N, Guertin MC, Turgeon J, Phillips MS, Rouleau JL, Tardif JC, White M; CANDIID II investigators. A prospective study of the impact of AGTR1 A1166C on the effects of candesartan in patients with heart failure. Pharmacogenomics. 2018 May;19(7):599-612. doi: 10.2217/pgs-2018-0004. Epub 2018 Apr 27. PMID 29701105